CLINICAL TRIAL: NCT00001210
Title: Prediction and Testing of Antigenic Sites of the AIDS Virus, HTLV-III Recognized by T Lymphocytes for the Development of Synthetic Vaccines
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 860199; 86-C-0199
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-10

CONDITIONS: HIV Infections; Healthy
Keywords: Blood Donors; Epitopes; HIV
MeSH Terms: conditions — HIV Infections

SUMMARY:
Subjects are healthy adult volunteers either at high risk for HIV infection or already known to be seropositive, who will donate blood for in vitro tests of T-cell function and in vitro responses to synthetic peptides corresponding to sequences from HIV proteins.

DETAILED DESCRIPTION:
Subjects are healthy adult volunteers either at high risk for HIV infection or already known to be seropositive, who will donate blood for in vitro tests of T-cell function and in vitro responses to synthetic peptides corresponding to sequences from HIV proteins.

ELIGIBILITY:
Inclusion criteria for the at risk group will be a statement from the donor that he is an active homosexual or bisexual.

Homosexual donors must not have AIDS.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1986-11; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Clerici M, Stocks NI, Zajac RA, Boswell RN, Bernstein DC, Mann DL, Shearer GM, Berzofsky JA. Interleukin-2 production used to detect antigenic peptide recognition by T-helper lymphocytes from asymptomatic HIV-seropositive individuals. Nature. 1989 Jun 1;339(6223):383-5. doi: 10.1038/339383a0. PMID 2524668
- [Background] Clerici M, Lucey DR, Berzofsky JA, Pinto LA, Wynn TA, Blatt SP, Dolan MJ, Hendrix CW, Wolf SF, Shearer GM. Restoration of HIV-specific cell-mediated immune responses by interleukin-12 in vitro. Science. 1993 Dec 10;262(5140):1721-4. doi: 10.1126/science.7903123.
- [Background] Pinto LA, Sullivan J, Berzofsky JA, Clerici M, Kessler HA, Landay AL, Shearer GM. ENV-specific cytotoxic T lymphocyte responses in HIV seronegative health care workers occupationally exposed to HIV-contaminated body fluids. J Clin Invest. 1995 Aug;96(2):867-76. doi: 10.1172/JCI118133. PMID 7635981